CLINICAL TRIAL: NCT02007876
Title: Mobility and Activity Training (MAT) to Optimize Outcomes for Older Adult Abdominal Surgery Patients
Acronym: MAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Michael Englesbe, Principal Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00062864
Record Dates: First submitted 2013-10-31; First posted 2013-12-11 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Gastrointestinal Malignancy
Keywords: Mobility; Activity; Training; Abdominal; Surgery; Adult
MeSH Terms: conditions — Motor Activity | interventions — Range of Motion, Articular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mobility and Activity Training (Experimental): Pre-operative: Participants will receive weekly sessions of higher level, task-specific transfer training. All MAT participants will learn the GCS set of exercises chosen to activate core muscles and lessen decline in core strength. These sessions will be supplemented by a home-based walking and physical activity enhancement program of the participants' choosing, focusing on attaining a safe community-based rate of perceived exertion. A pedometer and home exercise log will be used to encourage compliance and advance activities.
  Post-operative: Participants will be screened by physical therapy for standard physical therapy with focus on early mobilization. The GCS exercises taught pre-operatively will be reinstituted.
  Post-discharge/home: Participants will continue the GCS program and begin to return to elements of their pre-operative home-based MAT program. The program physical therapist will call weekly to review progress.
  Interventions: Behavioral: Mobility and Activity Training
- Normal activity (No Intervention): Pre-operative: Participants will be given the National Institute on Aging guide to home-based exercise but no further instruction or incentive for walking or physical activity enhancement.
  Post-operative: Participants will be screened by in-hospital physical therapy for standard physical therapy with focus on early mobilization. Those who do not receive physical therapy will not be given any additional training, as is standard for reimbursed hospital services.
  Post-discharge: Program nurse will call weekly to provide health education but no instruction or incentives for mobility or physical activity enhancement.

INTERVENTIONS:
Behavioral: Mobility and Activity Training — Pre-operative: Transfer training: bed and chair transferring exercises rising with and without use of hand assistance including supine to sit in or to the side in bed, and sit to stand from a normal and low height chair. GCS exercises: 1) supine pelvic bracing with transverse abdominal recruitment 2) hip bridges with abductor squeeze 3) supine bent leg abduction with light theraband and 4) supine isometric core and pelvic stabilization with legs flexed and shoulder flexion to raise arms over head with advancement to using theraband. For patients able to stand safely 5) standing mini squats against the wall.
  Post-operative: Early mobilization to include standard physical therapy techniques to enhance bed mobility, facilitated sit to stand and walking with therapist assist as needed. All GCS exercises begin 24 hr post op with goal of 5-10 reps and progressing to 3 sets of 10 reps. Participants will be encouraged to move from a roll to the side first supine to sit strategy by week 2.
  Arms: Mobility and Activity Training

SUMMARY:
In this pilot study a group of older adults undergoing midline laparotomy for gastrointestinal malignancy will participate in a mobility and activity training (MAT) program. MAT is designed to advance functional mobility and physical activity and spans the pre-operative, inpatient, and post-operative period. Patients undergoing abdominal surgery will be randomized to MAT versus control usual care and evaluated at their first appointment 4 weeks preoperatively (baseline), immediately prior to surgery, on hospital discharge, and 6 weeks post operatively. We hope to prove that abdominal surgery patients undergoing MAT will show less decline and earlier recovery in functional activity, and trunk and thigh muscle strength mass. This study is uniquely innovative in that it links functional activity assessment and training and analysis of trunk morphomics (muscle mass) in exploring mechanisms of post-operative recovery. Results from this pilot will be used to determine an effect size for the recruitment of a larger cohort and to study key surgical outcomes, including surgical complications, operative symptoms, hospital length of stay, and cost of care.

DETAILED DESCRIPTION:
Older and sicker patients are at increased risk of poor surgical outcomes, with more complications, longer lengths of stay, more utilization of skilled nursing facilities, increased mortality, and high costs when compared with younger and healthier patients undergoing similar procedures. In addition, more high-risk patients are having surgery, as overall surgical volumes are predicted to increase up to 47% (from 2000 to 2020). Within this context, efforts to improve surgical quality among high-risk patients have become of paramount importance and new proven strategies to improve surgical outcomes are needed.

Work by the PI Englesbe suggests that trunk muscle lean mass is strongly associated with poor surgical outcomes, suggesting an independent link between muscle loss (sarcopenia) and surgical outcome, even when controlling for comorbidity and functional impairment. Furthermore, their work notes that trunk muscle mass declines rapidly in the peri-operative period. Whether exercise interventions can remediate this risk is unknown. Few randomized control trials exist that address whether pre-operative exercise interventions can alter eventual post-operative outcomes, and none focus on training the trunk musculature in abdominal surgery patients. Further, trunk musculature is critical for mobilization and several published trials (such as in an intensive care unit) suggest that early mobilization is associated with improved outcomes. Thus, the link between reduction in muscle loss via exercise and improved mobility in post-surgical patients remains to be proven but seems promising. Co-PI Alexander has extensive experience in studies of mobility task assessment and enhancement in able and disabled adults. Of particular relevance to the present proposal are studies of rising from a bed (supine to sit) and from a chair (sit to stand) and the improvement that can be noted, using a task-specific approach in older adults at risk for mobility impairment. His most recent funded investigations focus on home-based mobility and physical activity enhancement.

We propose to pilot study a group of older adults undergoing midline laparotomy for gastrointestinal malignancy and who participate in a mobility and activity training (MAT) program. MAT is designed to advance functional mobility and physical activity and spans the pre-operative, inpatient, and post-operative period. Patients undergoing abdominal surgery will be randomized to MAT versus control usual care and evaluated at their first appointment 4 weeks preoperatively (baseline), immediately prior to surgery, on hospital discharge, and 6 weeks post operatively. We hope to prove that abdominal surgery patients undergoing MAT will show less decline and earlier recovery in functional activity, and trunk and thigh muscle strength mass. This study is uniquely innovative in that it links functional activity assessment and training and analysis of trunk morphomics (muscle mass) in exploring mechanisms of post-operative recovery. Results from this pilot will be used to determine an effect size for the recruitment of a larger cohort and to study key surgical outcomes, including surgical complications, operative symptoms, hospital length of stay, and cost of care.

Primary Aim 1: To determine the changes in extent of decline and in recovery of functional activity, strength, and muscle mass resulting from activity training (MAT) Primary hypothesis: Abdominal surgery patients randomized to MAT, as opposed to usual care controls (UC) and compared to their baseline evaluation 4 weeks pre-operatively, will have reduced loss of functional activity and reduced loss of muscle strength and mass in the trunk and thigh 6 weeks post-operatively.

Secondary Aim 1: To determine the effects of individual MAT program segments provided pre-operatively, in-hospital, and post-hospital discharge Secondary hypothesis: Abdominal surgery patients randomized to MAT, as opposed to UC, will have reduced loss of functional activity and reduced loss of muscle strength and mass in the trunk and thigh when comparing 1) baseline versus surgical admission; 2) surgical admission versus hospital discharge; and 3) hospital discharge versus post-operative follow-up at 6 weeks.

Exploratory Aim: To determine the effect of MAT on surgical complications, operative symptoms, hospital length of stay and peri-operative cost.

Exploratory hypothesis: Abdominal surgery patients randomized to peri-operative MAT, as opposed to UC, will have reduced surgical complications, fewer operative symptoms, shorter hospital length of stay, and lower cost of care.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparotomy for GI malignancy (colon resection, pancreatic resection, hepatectomy, resection of the bile ducts)
* Complete surgical resection (surgery on presumed cancer considered resectable by the attending surgeon.

Exclusion Criteria:

* Presumed benign disease as the indication for surgical resection.
* Received neo-adjuvant chemotherapy or radiation.
* Having preoperative severe hypo-albuminemia (albumin less than 3.0 g/dL).
* Having a previous ventral hernia repair or abdominal wall reconstruction.
* Morbid obesity (BMI>40)
* Participating in intensive (30 min per day) aerobic exercise program three times per week.
* Ongoing physical therapy in a relevant area (e.g. leg strengthening, balance and gait training)
* Myocardial infarction < 1 month
* Active symptoms of heart failure (NYHA grade II or higher)
* Atrial fibrillation with poor rate control (particularly during exercise) or high grade AV block
* Symptomatic obstructive valvular disease (primarily during exercise)
* Significant COPD
* Brittle diabetes (type I diabetes or multiple hypoglycemic episodes requiring assistance)
* Significant anemia (Hgb<7.0)
* Substantial dementia (Folstein Mini Mental State Examination <24 our of 30)
* Blood tests suggesting severe renal impairment (Cr>3.0)
* Alcohol intake >3oz/day
* Hemiplegia or lower limb amputation
* Acute medical conditions, such as acute flare-up of joint condition or infection
* Significant orthopedic or musculoskeletal condition that limits weight bearing activities
* Chronic pain syndrome affecting truncal areas (e.g. fibromyalgia)
* Unable to safely stand and walk, either with or without an assistive device

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Functional Activity and Strength | 10 weeks
  Participants randomized to MAT, as opposed to usual care controls (UC), will undergo physical therapy training as described in the intervention arm. The physical therapy will be used to assess functional activity and strength. Patients randomized into the MAT group will be compared to their baseline evaluation 4 weeks pre-operatively and the patients randomized into the UC group. We predict MAT study participants will have reduced loss of functional activity and reduced loss of muscle strength 6 weeks post-operatively.
Muscle Mass | 10 weeks
  Abdominal surgery patients will undergo 3-4 CT scans at baseline, pre-operatively, at hospital discharge, and at 6 weeks post-operatively. The CT scans will be used to measure changes in muscle mass. We predict MAT study participants will have reduced loss of muscle strength and mass in the trunk and thigh 6 weeks post-operatively.

SECONDARY OUTCOMES:
Effects of Individual MAT Program Segment | 10 weeks
  We hope to determine the effects of the individual MAT program segments provided pre-operatively, in-hospital, and at post-hospital discharge. Using the CT scans and physical therapy training and assessments, we will compare muscle mass and strength between each individual segment of the program. We predict that abdominal surgery patients randomized to MAT, as opposed to UC, will have reduced loss of functional activity and reduced loss of muscle strength and mass in the trunk and thigh when comparing 1) baseline versus surgical admission; 2) surgical admission versus hospital discharge; and 3) hospital discharge versus post-operative follow-up at 6 weeks.

OTHER OUTCOMES:
Effect of MAT on Surgical Complications | 6 weeks
  An additional exploratory aim of this study is to determine the effect of MAT on surgical complications. We predict that abdominal surgery patients randomized to peri-operative MAT, as opposed to UC, will have reduced surgical complications.
Effect of MAT on Cost of Care | 6 weeks
  An additional exploratory aim of this study is to determine the effect of MAT on peri-operative cost. We predict that abdominal surgery patients randomized to peri-operative MAT, as opposed to UC, will have lower cost of care
Effect of MAT of Operative Symptoms | 6 weeks
  An additional exploratory aim of this study is to determine the effect of MAT on operative symptoms. We predict that abdominal surgery patients randomized to peri-operative MAT, as opposed to UC, will have fewer operative symptoms.
Effect of MAT of Hospital Length of Stay | 6 weeks
  An additional exploratory aim of this study is to determine the effect of MAT on hospital length of stay. We predict that abdominal surgery patients randomized to peri-operative MAT, as opposed to UC, will have shorter hospital length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Englesbe, MD, Principal Investigator — University of Michigan; Neil Alexander, MD, Principal Investigator — University of Michigan; Angela E Thelen, BS, Study Director — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan-Mobility Research Center, Ann Arbor, Michigan
  - University of Michigan-Taubman Center, Ann Arbor, Michigan